CLINICAL TRIAL: NCT02827240
Title: A Peer Educator-delivered HIV Self-testing Intervention for Female Sex Workers in Zambian Border Towns
Brief Title: Zambian Peer-Educators for HIV Self-Testing Study
Acronym: ZEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: John Snow, Inc. (Industry); International Initiative for Impact Evaluation (Other)
Responsible Party: Principal Investigator, Till Barnighausen, Associate Professor, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 7041968-01
Record Dates: First submitted 2016-06-30; First posted 2016-07-11 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: HIV Infection
Keywords: Female sex workers; HIV testing; HIV self-test
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Direct Distribution (Experimental): The direct distribution arm consists of peer educators directly distributing HIV self-test kits to participants. Peer educators will briefly describe HIV self-testing to participants but will not provide extensive training on the use of the test kit. Peer educators also provide referral to existing services for HIV testing.
  Interventions: Other: Oral HIV Self-Testing
- Fixed Distribution (Experimental): The fixed distribution arm consists of peer educators distributing coupons to participants. The participants can then use the coupon to collect an HIV self-test kit at a participating distribution point, including drug stores, pharmacies, and health posts. Peer educators will briefly describe HIV self-testing to participants but will not provide extensive training on the use of the test kit. Peer educators also provide referral to existing services for HIV testing.
  Interventions: Other: Oral HIV Self-Testing
- Referral to Existing Services (No Intervention): Peer educators will not provide HIV self-tests to participants. Peer educators will only provide referral to existing services for HIV testing.

INTERVENTIONS:
Other: Oral HIV Self-Testing — The Oral HIV Self-Test is an in-home test that uses an oral swab to collect samples of oral mucosa that is used to detect the presence of HIV antibodies. The test is read after 20 minutes by the user. The test can be done by an individual at any time and place of the user's choosing. The test is read visually.
  Other Names: OraQuick HIV Self-Test
  Arms: Direct Distribution; Fixed Distribution

SUMMARY:
ZEST is a cluster-randomized trial designed to determine whether HIV self-tests are acceptable and improve HIV testing rates and HIV status knowledge among female sex workers in Zambian transit towns. This study will determine whether directly giving participants an HIV self-test or giving them a coupon to collect a test at a drug store or clinic improves outcomes compared to standard of care.

DETAILED DESCRIPTION:
Although Zambia has a generalized HIV epidemic, with approximately 13.3% of adults aged 15 to 49 living with HIV, the epidemic remains even more highly concentrated in key populations, including female sex workers (FSW). A particular concern for FSW is access to healthcare services, including HIV testing services. FSW face significant barriers to accessing healthcare. In other settings, evidence has suggested that stigma is a significant barrier to FSW seeking HIV testing. It is likely that similar mechanisms exist in Zambia. Evidence from Zambia has indicated that complex multilevel factors, such as stigmatization and harassment, contribute to vulnerability among FSW. User-controlled HIV prevention interventions that lead to empowerment of FSW may therefore be a powerful way to address the HIV epidemic in this key population.

Oral HIV self-testing consists of an oral swab kit that allows individuals to test for HIV in the privacy of their own homes whenever they want. The ease of use of HIV self-testing, that it can be done at any time, and that is completely private may make it an attractive alternative to currently-available HIV testing mechanisms for FSW in Zambia. HIV self-testing has generally been shown to be acceptable in a variety of populations, however evidence related to its uptake and acceptability remain sparse, especially among key populations and in Sub-Saharan Africa. This research will provide rigorous evidence of the uptake and efficacy of HIV self-testing for this population.

ZEST was designed to determine whether either direct distribution of HIV self-test kits via peer educators or distribution of HIV self-tests via coupons that participants can use to collect kits at collection points such as drug stores or health posts leads to better coverage of HIV testing and better awareness of HIV status. ZEST is a cluster-randomized trial in which peer educators recruit a small group of FSW participants, and the peer educator group is randomized to one of three study arms: 1) direct distribution of test kits, 2) fixed distribution of test kits, or 3) referral to standard of care HIV testing. The primary outcome is HIV testing in the past month measured at one and four months after the first peer educator visit (when the test kits or coupons are distributed in the intervention arms).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Female sex
* Reports exchanging sex (including vaginal, anal, and/or oral) for money or goods at least once in the past month
* Self-reported HIV negative with last HIV test at least 3 months OR HIV status unknown
* Permanent residence in the study town of enrollment (Kapiri, Livingstone, or Chirundu)
* Willing to be visited by and meet with assigned peer educator on a monthly basis over the 4-month study period

Exclusion Criteria:

* Less than 18 years of age on the enrollment date
* Has not exchanged any form of sex in the past one month
* Self-reported to be living with HIV
* Self-reported HIV negative status and tested within the past 3 months
* Living in PopART catchment area (Livingstone only)
* Concurrently participating in another HIV prevention study
* Meets criteria but does not wish to participate
* Other

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 965 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
HIV testing in the previous month | One month from first intervention visit
HIV testing in the previous month | Four months from first intervention visit

SECONDARY OUTCOMES:
Correct knowledge of HIV status | Four months from first intervention visit
HIV self-test kit use in the two intervention arms | One month from first intervention visit
HIV self-test kit use in the two intervention arms | Four months from first intervention visit
  In the intervention arms
Linkage to HIV care and confirmatory testing | One month from first intervention visit
Linkage to HIV care and confirmatory testing | Four months from first intervention visit
HIV risk perception and beliefs about acquiring HIV | One month from first intervention visit
HIV risk perception and beliefs about acquiring HIV | Four months from first intervention visit
HIV disclosure with sexual partners | One month from first intervention visit
HIV disclosure with sexual partners | Four months from first intervention visit
Condom use with commercial sexual partners since last visit | One month from first intervention visit
Condom use with commercial sexual partners since last visit | Four months from first intervention visit
Condom use with non-commercial sexual partners since last visit | One month from first intervention visit
Condom use with non-commercial sexual partners since last visit | Four months from first intervention visit
Average number of commercial sexual partners | One month from first intervention visit
Average number of commercial sexual partners | Four months from first intervention visit
Average number of non-commercial sexual partners | One month from first intervention visit
Average number of non-commercial sexual partners | Four months from first intervention visit
Intimate partner violence, including sexual, physical, or verbal | One month from first intervention visit
Intimate partner violence, including sexual, physical, or verbal | Four months from first intervention visit
HIV fatalism | One month from first intervention visit
HIV fatalism | Four months from first intervention visit
Self-reported self-efficacy as measured by the General Self Efficacy Scale | One month from first intervention visit
Self-reported self-efficacy as measured by the General Self Efficacy Scale | Four months from first intervention visit
Female sex worker empowerment as measured by Beattie et al 2014 | One month from first intervention visit
Female sex worker empowerment as measured by Beattie et al 2014 | Four months from first intervention visit
Pre-exposure prophylaxis preferences | One month from first intervention visit

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Oldenburg, ScD, MPH, Study Director — Harvard School of Public Health (HSPH); Till Baernighausen, MD, ScD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (3):
- Zambia (3):
  - John Snow, Inc, Lusaka, Livingstone
  - John Snow, Inc, Chirundu
  - John Snow, Inc, Kapiri

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available via International Initiative for Impact Evaluation's public access data repository.

REFERENCES:
- [Derived] Harling G, Chanda MM, Ortblad KF, Mwale M, Chongo S, Kanchele C, Kamungoma N, Barresi LG, Barnighausen T, Oldenburg CE. The influence of interviewers on survey responses among female sex workers in Zambia. BMC Med Res Methodol. 2019 Mar 15;19(1):60. doi: 10.1186/s12874-019-0703-2. PMID 30876402
- [Derived] Ortblad KF, Chanda MM, Musoke DK, Ngabirano T, Mwale M, Nakitende A, Chongo S, Kamungoma N, Kanchele C, Barnighausen T, Oldenburg CE. Acceptability of HIV self-testing to support pre-exposure prophylaxis among female sex workers in Uganda and Zambia: results from two randomized controlled trials. BMC Infect Dis. 2018 Oct 4;18(1):503. doi: 10.1186/s12879-018-3415-z. PMID 30286737
- [Derived] Oldenburg CE, Chanda MM, Ortblad KF, Mwale M, Chongo S, Kamungoma N, Kanchele C, Fullem A, Moe C, Barresi LG, Harling GD, Barnighausen T. Effect of HIV self-testing on the number of sexual partners among female sex workers in Zambia. AIDS. 2018 Mar 13;32(5):645-652. doi: 10.1097/QAD.0000000000001740. PMID 29494424
- [Derived] Chanda MM, Ortblad KF, Mwale M, Chongo S, Kanchele C, Kamungoma N, Fullem A, Dunn C, Barresi LG, Harling G, Barnighausen T, Oldenburg CE. HIV self-testing among female sex workers in Zambia: A cluster randomized controlled trial. PLoS Med. 2017 Nov 21;14(11):e1002442. doi: 10.1371/journal.pmed.1002442. eCollection 2017 Nov. PMID 29161260
- [Derived] Oldenburg CE, Ortblad KF, Chanda MM, Mwanda K, Nicodemus W, Sikaundi R, Fullem A, Barresi LG, Harling G, Barnighausen T. Zambian Peer Educators for HIV Self-Testing (ZEST) study: rationale and design of a cluster randomised trial of HIV self-testing among female sex workers in Zambia. BMJ Open. 2017 Apr 20;7(4):e014780. doi: 10.1136/bmjopen-2016-014780. PMID 28428187